CLINICAL TRIAL: NCT00826033
Title: Fluorine-18-α-Methyltyrosine Positron Emission Tomography to Measure Therapy
Brief Title: Fluorine-18-α-Methyltyrosine Positron Emission Tomography (18F-FMT PET) for Therapy Response in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Gunma University (Other)
Collaborators: J~pharma (Industry)
Other Study IDs: Mol Imaing 1
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Fluorine-18-α-methyltyrosine; Positron emission tomography; Lung cancer; chemotherapy; monitoring
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Therapy monitoring

SUMMARY:
L-[3-18F]-α-methyltyrosine (18F-FMT) is an amino-acid tracer for positron emission tomography (PET). The investigators evaluated the value of 18F-FMT PET for the assessment of therapy response in patients with lung cancer as compared with that of 2-[18F]-fluoro-2-deoxy-D-glucose (18F-FDG) PET.

The patients with lung cancer underwent PET studies with 18F-FDG and 18F-FMT before and after radio-/chemotherapy. The investigators used the ratio of the SUVmax of the mediastinal (N2) lymph node to the SUVmax of the primary tumor (N/P ratio ). All patients were divided into two groups of N/P ratio<1 and N/P ratio≥1, and the survival time was estimated by Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* primary lung cancer All patients received first-line chemotherapy

Exclusion Criteria:

* Patients with diabetus mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted at the Gunma University Hospital.
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Gunma University Graduate School of Medicine, Gunma, Japan